CLINICAL TRIAL: NCT02422914
Title: Benefits of Tobacco Free Cigarette Among Heavy Smokers Undergoing a Lung Cancer Screening Program: a Randomized Controlled Study
Brief Title: Benefits of Tobacco Free Cigarette
Acronym: BETOFREE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Collaborators: Fondazione Umberto Veronesi (Other); European Institute of Oncology (Other)
Responsible Party: Principal Investigator, claudio lucchiari, Prof, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R6314
Record Dates: First submitted 2015-01-14; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-01

CONDITIONS: Cigarette Smoking; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nicotine (Experimental): Smoking cessation program TFC and activity tracker. Three months low intensity counselling at distance program. Subject will also undergo a 3-months TFC (with nicotine) program; subjects smoking behaviour and wellbeing will be assessed at baseline, at 6 months and at one year. Life style will be evaluted by the use of an activity tracker and ad-hoc items.
  Interventions: Behavioral: Smoking cessation program TFC and activity tracker
- Nicotine-free (Placebo Comparator): Smoking cessation program TFC-free and activity tracker. Three months low intensity counselling at distance program. Subject will also undergo a 3-months TFC (nicotine-free) program; subjects smoking behaviour and wellbeing will be assessed at baseline, at 6 months and at one year. Life style will be evaluted by the use of an activity trackerand ad-hoc items.
  Interventions: Behavioral: Smoking cessation program TFC-free and activity tracker
- No-cig (Active Comparator): Smoking cessation program and activity tracker. Three months low intensity counselling at distance program;subjects smoking behaviour and wellbeing will be assessed at baseline, at 6 months and at one year. Life style will be evaluted by the use of an activity tracker and ad-hoc items.
  Interventions: Behavioral: Smoking cessation program and activity tracker

INTERVENTIONS:
Behavioral: Smoking cessation program TFC and activity tracker — Participants will receive a free TFC device and sufficient nicotine cartridges (8 mg/ml) to last the last of the procedure. Participants will be instructed to use the device ad libitum one week before their quit day (to be decided at the first contact) to familiarise themselves with its operation and on their designated quit day will stop smoking tobacco cigarettes and instead use the TFC exclusively for the next 11 weeks. The nicotine cartridges use will be monitored through the weekly diary and the monthly telephone. Lifestyle change will be monitored by the use of an activity tracker device (FitBit)
  Arms: Nicotine
Behavioral: Smoking cessation program TFC-free and activity tracker — Participants will receive a free TFC device and a set of 10 ml flacons enough to complete the trial. Participants will be instructed to use the device ad libitum one week before their quit day (to be decided at the first contact) to familiarise themselves with its operation and on their designated quit day will stop smoking tobacco cigarettes and instead use the TFC exclusively for the next 11 weeks.
  The actual use of the device and smoking habits will be monitored through the weekly diary and the monthly telephone. Lifestyle change will be monitored by the use of an activity tracker device (FitBit).
  Arms: Nicotine-free
Behavioral: Smoking cessation program and activity tracker — Participants undergo a motivational interview and low-intensity at distance counseling (the same counseling program of other groups) without any device.The actual smoking habits will be monitored through the weekly diary and the monthly telephone. Lifestyle change will be monitored by the use of an activity tracker device (FitBit).
  Arms: No-cig

SUMMARY:
Background. Smoking is considered a global public health problem. For this reason, the smoking dependence was called by experts as a global epidemic.

Over the past three years, this electronic devices (Tobacco Free Cigarettes, or TFC) has been an important expansion in many countries. Nevertheless, there is poor evidence that TFC are beneficial for smoking cessation. In particular, even though it has been proved that the nicotine replacement devices helps many individuals to give up smoking and to tolerate the withdrawal symptoms, it is still unclear their long-term effect. Hence, it must be tested its contribution in tobacco reduction. This protocol in particularly innovative, since it aims to test the efficacy of electronic devices in a screening program (the lung cancer prevention program COSMOS II at the IEO), where tobacco reduction is strictly needed in order to lower individual's risk.

Methods and Design. This experimental protocol has been designed with the main aim to investigate the role of Tobacco Free Cigarettes (TFC), also called e-cigarettes, in helping smokers to improve their lung health and to quit or reduce tobacco consuming. In particular, the investigators aim at investigating clinical (physical symptoms, with particular focus on breathing quality and difficulties), the behavioral (number of tobacco cigarettes smoked), and psychological (wellbeing, mood and quality of life) effects of shifting to TFC.

The investigators will also analyze, as a secondary aim, the psychological and lifestyle component of smokers involved in order to fine correlation data that might be used to compute a predictor index able to suggest the probability of success, with respect to the reduction of tobacco consuming, of the use of a TFC and to maintain the abstinence. The study will be organized as a nested randomized controlled study with two arms: one experimental group and one control group. The study will be nested in the screening program for lung cancer, where subjects will be recruited.

All subjects will be entered in a psycho-cognitive low-intensity counseling program (6 months), but in the experimental group a TFC (with or without nicotine) will be used as replacement device for three months, while in the control group only low-intensity counseling will be provided. Furthermore, a low-cost non-invasive electronic device (the FitBit activity tracker) will be used in order to monitor behavioral (lifestyle), sleep quality and physical activities.

DETAILED DESCRIPTION:
The World Health Organization has been estimated that cigarette smoking will claim the lives of 500 million people alive today and as many as one billion people in the 21st century. Even though clinical therapy for smoking cessation have showed efficacy, long-time abstinence rate is low yet.

Tobacco Free Cigarettes (TFC, also known as electronic cigarettes) are battery-operated devices designed to vaporize a liquid solution of propylene glycol and/or vegetable glycerin in which nicotine or other aromas may be dissolved.

The worth of these tools is that it reduces the risk for smoking related diseases. If the use of the TFC in heavy smokers favor a reduction of the cancers' risk, the role in antismoking program has not completed cleared yet. the World Health Organization (WHO) and the US Food and Drug Administration (FDA) have promoted the launch of research on this field.

In a prospective 6-month study, TFCs were shown to substantially decrease tobacco cigarettes consumption without causing significant side effects. The study showed that declines in cig/day use and expired carbon monoxide (CO) levels were observed at each study visits in all three study groups, with no consistent differences among study groups. Furthermore, rapid improvement of breathing symptoms were recorded.

However, tobacco cigarettes consumption after 1 year were reported only in about 10% of participants. This is probably due to the fact that the research was targeted to smokers non intended to quit. We argue that in motivated smokers much better result might be achieved.

From a physiological point of view TFCs appears to contrast craving for tobacco, in the same manner of a nicotine replacement therapy. In an overview of the Cochrane Library studies on 35.000 patients were assessed showing that the NRT utilization in antismoking treatment helps smokers in short-time (three months), but not in the long-time (six months). This is probably due to an exclusively focus on physiological issues.

The protocol provides the opportunity to test the efficacy of TFC tools in clinically controlled setting, in order to reduce tobacco consumption and improving clinical. Furthermore, the protocol is nested in the lung cancer screening program COSMOS II, that will allow subject recruitment and continuous monitoring. The Cosmos II (Continuous Observation of SMOking Subjects) aims to improve early diagnosis of lung cancer considered today as the most important life-saving tool. This is a Italian study, coordinated by IEO created to identify an optimal personalized protocol for early diagnosis in people subject to high risk of lung cancer. The COSMOS II will enroll 10,000 heavy smokers or former smokers throughout Italy. COSMOS II derives from the previous successful screening project COSMOS I.

Methods/Design

Main objectives:

To evaluate the impact of a three months TFC program to reduce smoking-related respiratory symptoms (dry cough, breath shortness, mouth irritation and catarrh) as consequence of a reduced tobacco cigarettes consumption among a CT screening population.

Secondary objectives:

1. To assess the success rate of smoking cessation attempts in the three groups 2 To monitor safety and toxicity during the study 3. To evaluate psychological and behavioral (lifestyle) effect of TFC 4. To assess the TFC use impact on quality of life .

More in details, the main aim of the project refers to the efficacy of TFCs in tobacco in improving the lung health of heavy smokers involved in the COSMOS II program. If proved safe and efficacy, TFC should be included in lung cancer screening programs as a standard tool to reduce the smoking-related risks for lung diseases. Naturally, this aim requires a scientific approach, since TFC should not increase the nicotine dependence. Another fundamental aim of the project refers to the efficacy of TFCs in tobacco consuming reduction. In particular, none study have already test the feasibility and the efficacy of these tools in limiting risk behaviors (tobacco smoking) among heavy smokers enrolled in a lung cancer screening program. Consequently, we want to analyze if providing TFC to participant in a controlled protocol will reduce tobacco consumption and related health problems and breathing problems. We also aim to analyse the psychological characteristics and needs of subjects enrolled in the COSMOS II program, in order to evaluate how risk perception (the premise of risk behaviour adoption) is associated with a psycho-cognitive profile. We argue that an important and successful screening project, as the COSMOS, should incorporate a comprehensive approach to the individual.

Finally, thanks to the use of a continuous data tracking system and the concomitant uses of questionnaire based anamnestic assessment of lifestyle and behavior habits, it will be possible to collect data in order to find consistency and discrepancies between the two methods.

TRIAL DURATION AND STUDY DESIGN

The project will last 24 months and is designed as a 6-months Nested Randomized Control Study and will be conducted in European Institute of Oncology.

The protocol addresses physical and clinical characteristics, in order to find out the effects of smokers' behavior, and psychological parameters, to test if some individual feature may hinder behavioral changes and the related positive effects on health. Indeed, heavy smokers are characterized by specific psycho-cognitive traits. In particulars, they generally present high level of impulsivity than non-smokers. At the same time, smoker tends to have an high level of activity in the behavioral approach system (BAS). It has been suggested that high BAS sensitivity is involved in addictive behaviors, for instance smoking. Individuals with high level of BAS are more incline to enact approaching behaviors and experience positive affect when they receive positive rewards. Furthermore, Dovratek and colleagues (2011) have demonstrated that smokers with high rumination attitude show a greater risk of relapse during the abstinence, especially, in those smokers characterized by high levels of impulsivity.

The experimental design, the timeline and nicotine doses were derived from previous research protocol that have demonstrated to be suited to achieve similar objectives. With respect to group 1 and group 2, a double blind randomization will be used, in order to avoid and confound effects. Consequently, participants using TFC won't know if the will "vape" nicotine-containing or nicotine-free.

Starting by this framework and In order to achieve the objectives described above we designed the protocol as follows:

1. To all subjects a physical, psychological, cognitive and behavioral (lifestyle) screening based on battery of fast and validated tools, will be administered. It will allow the assessment of the personality traits, the awareness's degree and the openness to change.
2. Each subject recruited will be involved in a behavioral support program (low-intensity counseling), in order to support subjects to track their data and to gather fast information when needed about the research activities.
3. The protocols will be organized in three arms:

   1. In the first arm subject will receive a 3-months TFC (with nicotine) program and a further 3-months monitoring program; they will undergo to a basal and final evaluation;
   2. In the second arm subject will receive a 3-months TFC (nicotine-free) program; they will undergo to a basal and final evaluation; they will be monitored for 6 month (data tracking);
   3. In the third arm, only baseline/final evaluation, data tracking and behavioral support will be delivered.

Subjects will be randomly assigned to each group after the first assessment point.

In each group, participants will follow a 6 month program (3 months of active program plus 3 months of monitoring). All participant will be monitored over the time for sleep quantity and quality of sleep and lifestyle, either through traditional instruments, and through the use of an electronic bracelet.

Participants will be trained to the use of the electronic bracelet and data will be collected through a cloud system allowing to compute statistical correlations between lifestyle, withdrawal symptoms, desire to smoke, recurrences, and so on. From this point of view, the research project will collect data currently not available. An e-messaging based helpline will be activated in order to offer full assistance to participants for the use of bracelets and research related activities.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects involved in the early lung cancer detection program (Cosmos II) of the European Institute of Oncology.
2. Subjects should have smoked at least 10 cigarettes a day for the past 10 years
3. Subjects that would like to reduce tobacco smoking but are not willing to be followed by a smoking center
4. To have an high motivational scoring (more than 10 points to the motivation questionnaire);
5. Signed informed consent

Exclusion Criteria:

1. symptomatic severe cardiovascular disease
2. symptomatic severe respiratory disease
3. regular psychotropic medication use
4. current or past history of alcohol abuse
5. use of smokeless tobacco or nicotine replacement therapy
6. pregnancy or breastfeeding.
7. Subjects involved in other antismoking program in the current year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary health (dry cough, breath shortness, mouth irritation) index | baseline, 6 months, 12 months
  To evaluate the impact of a three months TFC program to reduce smoking-related respiratory symptoms (dry cough, breath shortness, mouth irritation and catarrh) as consequence of a reduced tobacco cigarettes consumption among a CT screening population.

SECONDARY OUTCOMES:
Change in psychological wellbeing (had scale) | baseline, 6 months, 12 months
  To evaluate psychological and behavioral (lifestyle) effect of the TFC-based program
Change in number of daily cigarettes | baseline, 6 months, 12 months
  To assess the smoking behaviour within the three groups
Change in expired air carbon monoxide concentration | baseline, 6 months, 12 months
  To evaluate the impact of a three months TFC program to reduce smoking-related respiratory symptoms (dry cough, breath shortness, mouth irritation and catarrh) as consequence of a reduced tobacco cigarettes consumption among a CT screening population.
Change in values of the cough related quality of life questionnaire. | baseline, 6 months, 12 months
  To evaluate the impact of a three months TFC program to reduce smoking-related respiratory symptoms (dry cough, breath shortness, mouth irritation and catarrh) as consequence of a reduced tobacco cigarettes consumption among a CT screening population.
Change in daily activity (mean number of daily steps) | baseline, 6 months, 12 months
  To evaluate psychological and behavioral (lifestyle) effect of the TFC-based program
Change in lifstyle as measure by ad-hoc questionnaires | baseline, 6 months, 12 months
  To evaluate psychological and behavioral (lifestyle) effect of the TFC-based program

CONTACTS AND LOCATIONS:
Overall Officials: claudio lucchiari, PhD, Principal Investigator — University of Milan
Locations (1):
- University of Milan; European Institute of Oncology, Milan, Milan, Italy

REFERENCES:
- [Background] Bullen C, Howe C, Lin RB, Grigg M, Laugesen M, McRobbie H, Glover M, Walker N, Wallace-Bell M, Whittaker R, Rodgers A. Pre-cessation nicotine replacement therapy: pragmatic randomized trial. Addiction. 2010 Aug;105(8):1474-83. doi: 10.1111/j.1360-0443.2010.02989.x. Epub 2010 Jun 7. PMID 20528810
- [Background] Bullen C, Williman J, Howe C, Laugesen M, McRobbie H, Parag V, Walker N. Study protocol for a randomised controlled trial of electronic cigarettes versus nicotine patch for smoking cessation. BMC Public Health. 2013 Mar 8;13:210. doi: 10.1186/1471-2458-13-210. PMID 23496861
- [Background] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093
- [Background] Polosa R, Caponnetto P, Morjaria JB, Papale G, Campagna D, Russo C. Effect of an electronic nicotine delivery device (e-Cigarette) on smoking reduction and cessation: a prospective 6-month pilot study. BMC Public Health. 2011 Oct 11;11:786. doi: 10.1186/1471-2458-11-786. PMID 21989407
- [Background] Veronesi G, Bellomi M, Mulshine JL, Pelosi G, Scanagatta P, Paganelli G, Maisonneuve P, Preda L, Leo F, Bertolotti R, Solli P, Spaggiari L. Lung cancer screening with low-dose computed tomography: a non-invasive diagnostic protocol for baseline lung nodules. Lung Cancer. 2008 Sep;61(3):340-9. doi: 10.1016/j.lungcan.2008.01.001. Epub 2008 Mar 4. PMID 18308420
- [Derived] Lucchiari C, Masiero M, Veronesi G, Maisonneuve P, Spina S, Jemos C, Omodeo Sale E, Pravettoni G. Benefits of E-Cigarettes Among Heavy Smokers Undergoing a Lung Cancer Screening Program: Randomized Controlled Trial Protocol. JMIR Res Protoc. 2016 Feb 3;5(1):e21. doi: 10.2196/resprot.4805. PMID 26842790